CLINICAL TRIAL: NCT01177839
Title: Prospective, Hospital-based, Multicentre Study to Assess the Incidence of Intussusception in Children < 2 Years of Age in Singapore
Brief Title: Study to Assess the Incidence of Intussusception in Children < 2 Years of Age in Singapore
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 999910/193
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Intussusception
MeSH Terms: conditions — Intussusception

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Intussusception cohort: Subjects with Intussusception
  Interventions: Other: Screening sheets

INTERVENTIONS:
Other: Screening sheets — Reviewing screening sheets

SUMMARY:
This prospective study aims to estimate the incidence of intussusception among children < 2 years old through hospital-based surveillance in Singapore.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant aged < 24months at the time of diagnosis of intussusception.
* Subject is diagnosed with definite, probable, possible, suspected intussusception during the period of at least one year beginning at study start.
* Written informed consent obtained from the parent or guardian of the subject.

Exclusion Criteria:

* A male or female infant ≥ 24 months of age at the time of intussusception diagnosis.
* The subject has had a radiographically or surgically confirmed case of intussusception prior to the current episode.

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All subjects < 24 months of age seen on an in- or out-patient basis with a diagnosis of intussusception during at least a one year period beginning at study start.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2002-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of definite, probable and possible IS cases in children < 5 yrs of age | Average timeframe: one year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Singapore, Singapore

REFERENCES:
- [Derived] Phua KB, Lee BW, Quak SH, Jacobsen A, Teo H, Vadivelu-Pechai K, Gopala K, Liu Y. Incidence of intussusception in Singaporean children aged less than 2 years: a hospital-based prospective study. BMC Pediatr. 2013 Oct 8;13:161. doi: 10.1186/1471-2431-13-161. PMID 24103115